CLINICAL TRIAL: NCT03120234
Title: Comparison of Opioid Based and Opioid Free Anaesthesia in Transsphenoidal Surgery for Haemodynamic Stability and Recovery Characteristics
Brief Title: Comparison of Opioid Based and Opioid Free Anaesthesia in Transsphenoidal Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Post Graduate Institute of Medical Education and Research, Chandigarh (Other)
Responsible Party: Principal Investigator, Ayyawar Hareesh, principal investigator, Post Graduate Institute of Medical Education and Research, Chandigarh
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Health Services Research
Other Study IDs: MK/2950/MD/13121
Record Dates: First submitted 2017-01-06; First posted 2017-04-19 (Actual); Last update posted 2019-07-08 (Actual); Status verified 2019-07

CONDITIONS: Opioid Free Anaesthesia
MeSH Terms: interventions — Dexmedetomidine; Ketamine; Fentanyl

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Dexmedetomidine and ketamine (Experimental): The group will receive loading dose of dexmedetomidine 1mcg/kg over 10 Min followed by a maintenance of 0.5 mcg/ kg/ hr.ketamine 0.5 mg/kg will be given as bolus at the time of induction.
  Interventions: Drug: Dexmedetomidine; Drug: Ketamine
- fentanyl and placebo (Experimental): pts will receive fentanyl 2mcg/kg as bolus over 10 Mon followed by 1 mcg/ kg/hr as maintenance, instead of ketamine placebo(0.9%saline ) will be given in control group
  Interventions: Drug: Fentanyl; Drug: Placebos

INTERVENTIONS:
Drug: Dexmedetomidine
  Arms: Dexmedetomidine and ketamine
Drug: Ketamine
  Arms: Dexmedetomidine and ketamine
Drug: Fentanyl
  Arms: fentanyl and placebo
Drug: Placebos — o.9% normal saline will be used instead of ketamine
  Arms: fentanyl and placebo

SUMMARY:
This study has been planned to compare the effect of opioid free anaesthesia using dexmedetomidine and ketamine with opioid based anaesthesia using fentanyl in maintaining the intraoperative hemodynamic stability and recovery characteristics in patients undergoing Transsphenoidal surgery of pituitary tumors.

DETAILED DESCRIPTION:
Opioid Free Anesthesia (OFA) is a technique where no intraoperative opioid is administered during the anesthetic management. Opioid free anesthesia is usually achieved through sympatholysis, analgesia, and anesthesia with dexmedetomidine and analgesia with low dose ketamine. In addition paracetamol and other non-steroidal anti inflammatory drugs (NSAIDS) may be used as adjuncts to the multi-modal pain regimen.

Dexmedetomidine, a highly selective agonist of the alpha2 adrenergic receptor, has many clinical benefits, such as sedation, analgesia, preventing unwanted stress responses and low risk of respiratory depression. Because of concern that opioids might cause perioperative respiratory depression, substitution with dexmedetomidine will be helpful with its analgesic and sympatholytic properties. Dexmedetomidine has shown to reduce minimum alveolar concentration (MAC) of inhalational anesthetics and the requirement of perioperative opioid by 30-50%. In neurosurgical patients, dexmedetomidine is helpful in maintaining intracranial pressure (ICP) and intraoperative hemodynamic stability, especially during intubation and extubation. It can allow for faster awakening and thus an earlier neurological examination by decreasing necessary volatile agent and opioid doses.

Ketamine, an N-methyl-d-aspartate(NMDA) antagonist, blunts central pain sensitization at sub-anesthetic doses (0.5 mg/kg or less) and has been studied extensively as an adjunct for perioperative analgesia. Sub-anesthetic ketamine improves pain scores and reduces perioperative opioid consumption in a broad range of surgical procedures.Recent literature has suggested that adjuvant ketamine administration in mechanically ventilated patients has no cerebrovascular effects.

The present study has been planned to compare the effect of opioid free anesthesia using dexmedetomidine and ketamine with opioid based anesthesia using fentanyl in maintaining the intraoperative hemodynamic stability and recovery characteristics in patients undergoing TSS of pituitary tumors.

ELIGIBILITY:
Inclusion Criteria:

* patients suffering significant pituitary adenocarcinomas posted for transsphenoidal resection of tumor
* age group between 18 to 65 yr
* Both males and females
* ASA physical status 1 to 2

Exclusion Criteria:

* pts taking opioid for chronic pain
* Pregnant or nursing woman
* Preoperative GCS <15
* HR<50/min
* Patients with allergies to study medication
* Patients with psychiatric disorder
* Patients with unstable cardiorespiratory disorder
* Patients with hepatic and renal insufficiency

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2017-10 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
To measure the emerence and extubation times in both groups | 15minutes
  it is measured by noting the time for emergence and extubation after stopping inhalational anaesthesia.
to measure the level of emergence in both the groups | 15min
  using Riker sedation-agitation score
to measure the level of cognition in both the groups | 15min
  using Short orientation memory concentration test (SOMC test)

SECONDARY OUTCOMES:
comparison of intraoperative hemodynamic stability in both the groups | intra operative period
  this will be done by monitoring intraoperative hemodynamics and noting down no of events of hypotension and hypertension and noting down the rescue drug requirements.
postoperative pain assessment by using numeric rating scale | 24 hrs
comparing postoperative analgesic dose requirement in both the groups | 24hrs

CONTACTS AND LOCATIONS:
Overall Officials: AYYAWAR HAREESH, MBBS, Principal Investigator — Post Graduate Institute of Medical Education and Research, Chandigarh
Locations (1):
- Post graduation institute of medical education and research, Chandigarh, India

IPD SHARING:
Plan to Share IPD: Undecided